CLINICAL TRIAL: NCT00545675
Title: Multi-center, Double-blind, Randomized, Comparative Phase 4 Clinical Trial to Evaluate the Efficacy and Safety of Co-administration of Abilify and Depakote in 24-week Treatment of Mania in Patients With Bipolar Disorder Remitted After 6-week Treatment With Abilify and Depakote
Brief Title: Abilify in Bipolar Disorder for 24 Weeks Treatment Effectiveness
Acronym: SMART-M
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Yonghui Jeong, Clinical Research Manager, Korea Otsuka Pharmaceutical Co.,Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-KOB-0702
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2009-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Abilify(aripiprazole) + Depakote(divalproate)
  Interventions: Drug: Abilify(aripiprazole)
- 2 (Placebo Comparator): Divalproate + Placebo
  Interventions: Drug: Depakote (divalproate)

INTERVENTIONS:
Drug: Abilify(aripiprazole) — Abilify and Depakote in 24-week treatment of mania in patients with bipolar disorder
  Arms: 1
Drug: Depakote (divalproate) — Placebo and Depakote in 24-week treatment of mania in patients with bipolar disorder
  Arms: 2

SUMMARY:
To demonstrate the difference between Abilify with Depakote vs. Placebo with Depakote in 24-week treatment in patients with remission status after Abilify with Depakote in the 6-week study of acute mania in patients with bipolar disorder

DETAILED DESCRIPTION:
Further study details as provided by Korea OIAA

ELIGIBILITY:
Inclusion Criteria:

1. Mania or mixed episode of bipolar disorder according to DSM-IV
2. Male and female between the age of 18 and 65 (In case of child-bearing women, negative pregnancy test results should be confirmed before the administration of the investigational drug and appropriate contraception be used. Pregnant and breast-feeding women cannot be included)
3. Patients who can consent to participate in this clinical trial
4. Patients who understand this trial and comply with all protocol requirements
5. Patients who fulfill the following remission criteria for bipolar disorder in the two consecutive evaluation performed every week at Week 6 of 6-week study and thereafter:

(Definition of remission: a score less than 12 on the YMRS total score and simultaneously a score less than 13 on the MADRS total score)

Exclusion Criteria:

1. Patients with the following clinical symptoms diagnosed using DSM-1. Patients with the following clinical symptoms diagnosed using DSM-IV:

   * Delirium, dementia, amnestic or other cognitive disorders
   * Schizophrenia or schizoaffective disorder
2. Patients who do not respond to clozapine
3. Patients who are expected to require the administration of prohibited concomitant drugs during the clinical trial period
4. Patients diagnosed with substance-related disorder according to DSM-IV within the past 3 months (abuse, intoxication, dependency and/or withdrawal symptoms). The abuse of benzodiazepines is included with the exception of caffeine or nicotine.
5. Patients known to have allergy or hypersensitivity reaction to Abilify(aripiprazole) or other quinolinones
6. Patients at high risk of suicide attempt or with the history of murder or mental status test
7. Patients with the history of neuroleptic malignant syndrome
8. Patients with the past history which may cause serious adverse events that can affect the safety or efficacy evaluation during the clinical trial period
9. Patients with clinically significantly abnormal laboratory results, vital sign or ECG results
10. Pregnant women or child-bearing women who do not or cannot use appropriate contraception
11. Patients with the history of convulsive disorder
12. Patients judged to have decreased compliance to the investigational drugs during a 6-week trial period by an investigator
13. Patients who commit serious protocol violation during a 6-week trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Time to recurrence of bipolar disorder from randomization | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Won-Myong Bahk, MD, Principal Investigator — St Mary's Hospital, London
Locations (1):
- St. Mary's Hospital, Seoul, South Korea